CLINICAL TRIAL: NCT03349112
Title: The Effect of Lidocaine on Perceived Comfort and Swallowing Pressures During High Resolution Pharyngeal Manometry
Brief Title: Study: Manometry With & Without Lidocaine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015-0485; A539772 (Other: UW Madison); SMPH/SURGERY/SURGERY*SP (Other: UW Madison)
Record Dates: First submitted 2017-08-31; First posted 2017-11-21 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: Normal
Keywords: Manometry; Lidocaine; Pharyngeal; High Resolution Pharyngeal Manometry (HRPM); Pressure
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Intervention Model Description: During both the anesthetized and non-anesthetized conditions as per standard of care, the study team member will apply 1 mL of 2% viscous lidocaine to each nares prior to the passage of the catheter. During only the anesthetized condition, subjects will receive up to .8 ml of a 4% Lidocaine spray to both nares.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anesthetized (Active Comparator): A study team member will apply 1 mL of 2% viscous lidocaine to each nares prior to the passage of the catheter, Participants in this group will additionally receive .8 mL of a 4% Lidocaine spray to both nares prior to HRPM.
  Interventions: Behavioral: 4% Lidocaine Spray; Behavioral: 2% Viscous Lidocaine
- Non-Anesthetized (Placebo Comparator): A study team member will apply 1 mL of 2% viscous lidocaine to each nares prior to the passage of the catheter. Randomized participants in this group will not receive .8 mL of a 4% Lidocaine spray prior to HRPM .
  Interventions: Behavioral: 2% Viscous Lidocaine

INTERVENTIONS:
Behavioral: 4% Lidocaine Spray — 2% Viscous Lidocaine is applied to the nares as standard of care. In this intervention, 4% lidocaine spray is applied additionally.
  Arms: Anesthetized
Behavioral: 2% Viscous Lidocaine — 2% Viscous Lidocaine is applied to the nares as standard of care. This intervention is considered as the control group.

SUMMARY:
The purpose of this study is to determine whether subjects report a difference in comfort with High Resolution Pharyngeal Manometry (HRPM) conducted following application of lidocaine as an anesthetic as compared to HRPM conducted without anesthetic.

DETAILED DESCRIPTION:
High resolution pharyngeal manometry (HRPM) is used for assessing swallowing pressure along the length of the pharynx and upper esophageal sphincter. Pressure measurements in the region of the velopharynx, tongue base, and upper esophageal sphincter are obtained by passing a catheter with pressure sensors through the patient's nose and past the upper esophageal sphincter. Patients are presented various volumes of liquid to swallow and potentially asked to perform postural strategies such as a head turn or chin tuck during swallowing while the catheter is in place. Clinically, approximately 90% of patients report various discomfort associated with the procedure. Discomfort can result in patient refusal to participate or an inaccurate picture of a patient's swallowing pressures. Conversely, use of anesthesia can potentially alter swallowing physiology.

Recent studies have studied the effects of lidocaine on penetration/aspiration and subject discomfort during flexible endoscopic evaluations, yet findings are inconclusive or contradictive. Investigators aim to determine whether subjects report a difference in comfort with HRPM conducted following application of lidocaine as an anesthetic as compared to HRPM conducted without anesthetic.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female adults 18-65.
2. All races.
3. Able to consent for self.

Exclusion Criteria:

1. History of dysphagia.
2. History of previous pharyngeal or esophageal manometry.
3. History of facial fracture or abnormalities precluding passage of catheter through nares.
4. History of esophageal pathology including previous resection or perforation.
5. Pregnant
6. Known lidocaine allergy or sensitivity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-12-22 (Actual); Primary Completion 2018-11-09 (Actual); Study Completion 2018-11-09 (Actual)

PRIMARY OUTCOMES:
A quantifiable difference of perceived comfort reduction during HRPM with or without lidocaine as assessed through analysis of a visual analog scale. | Assessing the change of the visual analog scale between two procedural study visits. Data will be reported at study completion, an average of 1 year.
  Following HRPM without additional lidocaine and following HRPM with additional lidocaine, the subject will be asked to rate their level of comfort during the procedure using a visual analog scale.

CONTACTS AND LOCATIONS:
Overall Officials: Jodi Hernandez, MS, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin - Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No